CLINICAL TRIAL: NCT04351308
Title: A Randomized Trial of Comparison of MAPI+Camrelizumbab Verus API+Apatinib Versus MAPI in Patients With a Poor Response to Preoperative Chemotherapy for Newly Diagnosed High-grade Osteosarcomaies : an Open-label, Exploratory Study
Brief Title: Comparison of MAPI+Camrelizumab Versus API+Apatinib Versus MAPI in Patients With a Poor Response to Preoperative Chemotherapy for Newly Diagnosed High-grade Osteosarcoma
Acronym: MAPAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Chinese Sarcoma Study Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma 09
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Osteosarcoma; Survival; Chemotherapy Effect; Toxicity, Drug
Keywords: osteosarcoma; doxirubicin; cisplatin; methotrexate; ifosfamide; apatinib; camrelizumab
MeSH Terms: conditions — Osteosarcoma; Drug-Related Side Effects and Adverse Reactions | interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- API+apatinib (Experimental): AP = Doxorubicin (Adriamycin) 20 mg/m2/day * 2 day (total/cycle 40 mg/m²)
  + Cisplatin 100 mg/m2/course (total/cycle 120 mg/m²);
  I = Ifosfamide 2000 mg/m2/day *5 day (total/cycle 10000 mg/m²);
  apatinib = 500 mg QD;
  Interventions: Drug: MAPI chemotherapy; Drug: Apatinib Mesylate
- MAPI+camrelizumab (Experimental): AP = Doxorubicin (Adriamycin) 37.5 mg/m2/day * 2day (total/cycle 75 mg/m²)
  + Cisplatin 120 mg/m2/course (total/cycle 120 mg/m²);
  M = Methotrexate 12000 mg/m2 (total/cycle 12000 mg/m²) with leucovorin rescue;
  I = Ifosfamide 2400 mg/m2/day *5day (total/cycle 12000 mg/m²);
  camralizumab = 200mg ivgtt. Q2W;
  Interventions: Drug: MAPI chemotherapy; Drug: Camrelizumab
- MAPI (Active Comparator): AP = Doxorubicin (Adriamycin) 37.5 mg/m2/day * 2day (total/cycle 75 mg/m²)
  + Cisplatin 120 mg/m2/course (total/cycle 120 mg/m²);
  M = Methotrexate 12000 mg/m2 (total/cycle 12000 mg/m²) with leucovorin rescue;
  I = Ifosfamide 2400 mg/m2/day *5day (total/cycle 12000 mg/m²);
  Interventions: Drug: MAPI chemotherapy

INTERVENTIONS:
Drug: MAPI chemotherapy — AP = Doxorubicin (Adriamycin) 37.5 mg/m2/day * 2day (total/cycle 75 mg/m²)
  + Cisplatin 120 mg/m2/course (total/cycle 120 mg/m²) ; M = Methotrexate 12000 mg/m2 (total/cycle 12000 mg/m²) with leucovorin rescue; I = Ifosfamide 2400 mg/m2/day *5day (total/cycle 12000 mg/m²)
Drug: Apatinib Mesylate — anti-angiogenesis tyrosine kinase inhibitors 500 mg orally daily
  Arms: API+apatinib
Drug: Camrelizumab — anti-PD-1 antibody 200mg ivgtt. Q2W
  Arms: MAPI+camrelizumab

SUMMARY:
Treatment strategies for high-grade osteosarcoma with multidrug chemotherapy and resection result in 3-year event-free survival of 60-70%. The most common factors predicting survival are presence of metastases, histological response to preoperative chemotherapy and complete surgical resection. Four of the active drugs in osteosarcoma include cisplatin, doxorubicin, high-dose methotrexate and ifosfamide and this combination (MAPI), given preoperatively and postoperatively, is widely used for the treatment of osteosarcoma in China. Apatinib also has activity in advanced setting and when incorporated into the treatment of patients with metastatic disease seemed to improve progression-free survival. Combination of apatinib and camrelizumab resulted in durable therapuetic effect in selected cases. Though EURAMOUS-1 suggested that changing chemotherapy postoperatively on the basis of histological response did not improve outcomes. The exploratory study with radomised design to compare combination of chemotherapy with target drug or combination of chemotherapy with anti-PD-1 antibody versus standard chemotherapy has not been tried yet. Thus we aim to investigate the efficacy and toxicity of these combiantions versus standard chemotherapy in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade osteosarcoma, including second malignancies
* Tumor (primary, metastatic, or both) resectable OR is expected to become resectable after neoadjuvant induction chemotherapy
* Suitable for neoadjuvant chemotherapy and adjuvant chemotherapy
* Performance status - Lansky 50-100% (for patients under 16 years of age); Performance status - WHO or ECOG 0-2 with a life expectancy >3 months
* normal cardiac function (shortening fraction >28%), normal hearing, normal bone marrow as shown by an absolute neutrophil count of at least 1·5 × 10⁹ cells per L (or a white blood cell count of at least 3 × 10⁹ cells per L if neutrophil count is not available), and a platelet count of at least 100 000 platelets per μL
* Patients were also required to have a serum bilirubin concentration of at most less than 1·5 times the upper limit of normal and a normal creatinine concentration for their age as per protocol
* Women of child-bearing potential had to take adequate contraceptive measures and have a negative pregnancy test within 7 days of study entry.

Exclusion Criteria:

* patients who have recieved anti-angiogenic TKIs or anti-PD-1/PD-L1 antibodies
* allergy to chemotherapy or apatinib or camrelizumab
* other severe illness (eg, psychosis or previous history of cardiovascular disease)
* symptomatic or known CNS metastases
* previous or concurrent second primary malignant tumours
* had uncontrolled complications such as diabetes mellitus, coagulation disorders, urine protein ≥ ++, and so on
* had other infections or wounds
* pregnant or breastfeeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
event-free survival rate | 2 years
  from initial treatment after definitive surgery to progression/death/ last follow up

SECONDARY OUTCOMES:
overall survival rate | 5 years
  from initial treatment after definitive surgery to death/ last follow up

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, M.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China